CLINICAL TRIAL: NCT05827627
Title: Assessment of Efficacy of Two Different Simulation Techniques Used in Breech Birth Management Training: A Randomised Controlled Study
Brief Title: Simulation Techniques Used in Breech Birth Management Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Yasemin Hamlaci Baskaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 03052019
Record Dates: First submitted 2023-03-31; First posted 2023-04-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Breech Presentation
Keywords: breech birth; simulation; midwifery students; training
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Intervention Model Description: The study was conducted in two groups: a pelvic simulator group (PSG) and a computer-based simulator group (CBSG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic simulator group (PSG) (Other): The trainer positioned the foetus in the pelvic simulator in frank breech presentation. Descent of the baby in the pelvic simulator was administered by a person independent of the study and the training.
  Interventions: Other: simulation
- Computer-based simulator group (CBSG) (Experimental): The trainer positioned the foetus in the computer-based full-body childbirth simulator in frank breech presentation. The pregnancy simulator streamed audio to increase reality and the patient monitor displayed vital signs of the pregnant simulator and foetal heart rate.
  Interventions: Other: simulation

INTERVENTIONS:
Other: simulation — Midwifery student directing the birth of a fetus with frank breech presentation.

SUMMARY:
This study was conducted to assess the effect of two different simulation techniques that are used to improve breech birth management skills of midwifery students on the anxiety, self-efficacy, skill and knowledge levels of students.

DETAILED DESCRIPTION:
Professional midwives are an integral part of delivering quality sexual, reproductive, maternal, and newborn healthcare. Midwives must have the skills and knowledge to assist childbirth and identify problems when labour progresses well. When a midwife examines a woman in labour, she may encounter an unexpected breech presentation. Therefore, it is important for midwives to have the skills and knowledge to deliver breech babies and assist mother and baby. Recently, caesarean section has been preferred in breech presentations. However, if breech presentation is diagnosed after the active phase, there may not be enough time for preparations for caesarean section, or the woman may refuse surgical intervention. In both cases, the midwife who examines the woman should inform the obstetrician immediately and, if possible, seek the assistance of another midwife or physician who is experienced in vaginal breech delivery in the management of childbirth. This may result in foetal injury at the hands of inexperienced providers. Midwives and physicians providing intrapartum care must have good training on breech birth manoeuvres and management of the second phase in order to minimise complications. Furthermore, one of the competencies specified by the International Confederation of Midwives (ICM) in midwifery practices is to 'Undertake appropriate manoeuvres and use maternal position to facilitate vertex, face, or breech birth'. Many midwifery education programmes now use various simulators and simulation training to improve the skills of students in high-risk deliveries.

Simulation-based training is an educational method bridging theory and practice and is one of the preferred skill training methods at educational institutions for healthcare professionals. Reasons for preferring this method can be listed as: limited access of students to a qualified faculty in clinical settings, low frequency of situations and limited exposure to actual patients. There are also ethical reasons for using simulation in the education of students, such as minimising risks for patients and providing students with an opportunity to learn through simulation. Simulation training provided before clinical practice helps students to feel safe and well prepared for the clinical setting. Having repetitive training in a safe and secure environment without fear of comprising patient safety is viewed as important for students.

There has been growing interest in simulation and skill training in midwifery education. Simulation laboratories have been established at many universities and training hospitals. The most commonly used simulation types in midwifery education are scenario-based skill training with standardised patients, scenario-based high-technology simulators, and simulators not involving technological design (e.g., episiotomy simulators, pelvic simulators for childbirth, simulator dolls). In midwifery education, it is aimed to teach students basic and advanced practice skills, such as delivering a certain number of babies, making and repairing episiotomies and assisting breech births. Simulation-based learning develops professional competence in midwifery educators as well as equipping and empowering midwifery students regarding practices. In undergraduate midwifery education, students are provided with obstetric skill training in electronic foetal monitoring (EFM), childbirth management, shoulder dystocia, postpartum haemorrhage, breech birth, umbilical cord prolapse and perineal repair (laceration and episiotomy). It has been determined that simulation-based training affected positively participants' perceived readiness. Training provided with high-fidelity, high-technology simulators has been determined to enhance students' self-efficacy, confidence and satisfaction.

It has been aimed to find answers of "is there any difference in students' levels of anxiety, self-efficacy and knowledge on breech birth management between a pelvic simulator group and a computer-based simulator group before and after the training?" and "is there any difference in improving skills in breech birth management between the two groups?"

ELIGIBILITY:
Inclusion Criteria:

1. Students who were enrolled in the senior year
2. Students who participated in the High-Risk Birth Management course
3. Students who received theoretical information on breech birth management

3. Students who agreed to take part in the study

Exclusion Criteria:

1. Students who failed in the High-Risk Birth Management course
2. Students who did not participate in theoretical education of breech birth management

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory Score Change | pre-intervention, 1 hour after intervention
  The inventory, developed by Spielberger et al. (1970), is a self-evaluation questionnaire involving short evaluations (Spielberger et al., 1983). Its validity and reliability study in Turkey was conducted by Öner and Lecompte (1983) (Öner & Le Compte, 1983). The inventory consists of two different questionnaires with 40 items in total. The STAI consists of 20 items that aim to assess how the individual feels at a specific time under specific conditions by considering their present feelings and was used in our study. It is a 4-point Likert scale ranging from 'Not at all' to 'Very much so'. The maximum score that can be obtained from the scale is 80, and the minimum score is 20. Higher scores are correlated with higher levels of anxiety.
Self-Efficacy Scale Score Change | pre-intervention, 1 hour after intervention
  Developed by Sherer et al. (1982), the Self-Efficacy Scale is a 5-point Likert scale and consists of 23 items (Gözüm & Aksayan, 1999; Sherer et al., 1982). The scale measures generalised, non-specific perception of self-efficacy. The scores to be obtained from the scale range from 23 to 115; higher scores represent a good level of self-efficacy perception.
Breech Birth Management Information Form Score Change | pre-intervention, 1 hour after intervention
  This form was developed based on relevant literature (Marshall & Raynor, 2014; Posner et al., 2013; Shuttler, 2018; Walker, Reading, et al., 2017). It consisted of 17 statements intended to measure the students' level of knowledge on breech birth management. The statements were prepared to include eight correct and nine incorrect statements which were answered by the participants as 'I agree', 'I disagree' or 'I have no idea'. One point was awarded for correct answers and zero points for incorrect and 'no idea' answers. Higher knowledge scores denote a higher level of knowledge on breech birth management.
Breech Birth Management Skill Assessment Form | 1 hours
  The Breech Birth Management Skill Assessment Form was prepared by reviewing the relevant literature (Hardy et al., 2020; Jordan et al., 2016; Shuttler, 2018; Walker, Breslin, et al., 2017). The form consisted of 19 items involving steps of breech birth management, such as hand washing, protecting privacy, making necessary explanations to the pregnant woman, determining the presentation of the foetus, informing the pregnant woman about pushing and cooperating, waiting for the umbilical cord to be delivered, assisting the delivery of the baby's arm and head with suitable manoeuvres, informing the woman about the outcomes, and recording the procedures on an observation sheet.The score to be obtained from the form ranged from 19 to 57.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Başkaya, Study Director — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aggarwal R, Mytton OT, Derbrew M, Hananel D, Heydenburg M, Issenberg B, MacAulay C, Mancini ME, Morimoto T, Soper N, Ziv A, Reznick R. Training and simulation for patient safety. Qual Saf Health Care. 2010 Aug;19 Suppl 2:i34-43. doi: 10.1136/qshc.2009.038562. PMID 20693215
- [Result] Bogossian F, McKenna L, Higgins M, Benefer C, Brady S, Fox-Young S, Cooper S. Simulation based learning in Australian midwifery curricula: results of a national electronic survey. Women Birth. 2012 Jun;25(2):86-97. doi: 10.1016/j.wombi.2011.02.001. Epub 2011 Mar 8. PMID 21388902
- [Result] Bogren M, Rosengren J, Erlandsson K, Berg M. Build professional competence and Equip with strategies to empower midwifery students - An interview study evaluating a simulation-based learning course for midwifery educators in Bangladesh. Nurse Educ Pract. 2019 Feb;35:27-31. doi: 10.1016/j.nepr.2019.01.002. Epub 2019 Jan 10. PMID 30658269
- [Result] Carbillon L, Benbara A, Tigaizin A, Murtada R, Fermaut M, Belmaghni F, Bricou A, Boujenah J. Revisiting the management of term breech presentation: a proposal for overcoming some of the controversies. BMC Pregnancy Childbirth. 2020 May 3;20(1):263. doi: 10.1186/s12884-020-2831-4. PMID 32359354
- [Result] Deering S, Brown J, Hodor J, Satin AJ. Simulation training and resident performance of singleton vaginal breech delivery. Obstet Gynecol. 2006 Jan;107(1):86-9. doi: 10.1097/01.AOG.0000192168.48738.77. PMID 16394044
- [Result] Hardy L, Garratt JL, Crossley B, Copson S, Nathan E, Calvert K, Epee-Bekima M. A retrospective cohort study of the impact of In Time obstetric simulation training on management of vaginal breech deliveries. Aust N Z J Obstet Gynaecol. 2020 Oct;60(5):704-708. doi: 10.1111/ajo.13132. Epub 2020 Feb 17. PMID 32067227
- [Result] Hunter LA. Vaginal breech birth: can we move beyond the Term Breech Trial? J Midwifery Womens Health. 2014 May-Jun;59(3):320-7. doi: 10.1111/jmwh.12198. Epub 2014 Apr 24. PMID 24762034
- [Result] Jordan A, Antomarchi J, Bongain A, Tran A, Delotte J. Development and validation of an objective structured assessment of technical skill tool for the practice of breech presentation delivery. Arch Gynecol Obstet. 2016 Aug;294(2):327-32. doi: 10.1007/s00404-016-4063-4. Epub 2016 Mar 11. PMID 26969652
- [Result] Lendahls L, Oscarsson MG. Midwifery students' experiences of simulation- and skills training. Nurse Educ Today. 2017 Mar;50:12-16. doi: 10.1016/j.nedt.2016.12.005. Epub 2016 Dec 16. PMID 28006699
- [Result] Maskalova E, Urbanova E, Baskova M, Kvaltinyova E. Experience of lecturers with simulation training in midwifery education in Slovakia. Midwifery. 2018 Apr;59:1-3. doi: 10.1016/j.midw.2018.01.001. Epub 2018 Jan 5. PMID 29331775
- [Result] Stone H, Crane J, Johnston K, Craig C. Retention of Vaginal Breech Delivery Skills Taught in Simulation. J Obstet Gynaecol Can. 2018 Feb;40(2):205-210. doi: 10.1016/j.jogc.2017.06.029. Epub 2017 Aug 15. PMID 28821414
- [Result] Stoodley C, McKellar L, Steen M, Fleet J. Simulation in midwifery education: A descriptive explorative study exploring students' knowledge, confidence and skills in the care of the preterm neonate. Nurse Educ Pract. 2020 Jan;42:102635. doi: 10.1016/j.nepr.2019.102635. Epub 2019 Oct 10. PMID 31864035
- [Result] Tyer-Viola L, Zulu B, Maimbolwa M, Guarino A. Evaluation of the use of simulation with student midwives in Zambia. Int J Nurs Educ Scholarsh. 2012 Aug 9;9:/j/ijnes.2012.9.issue-1/1548-923X.2379/1548-923X.2379.xml. doi: 10.1515/1548-923X.2379. PMID 22947661
- [Result] Vermeulen J, Beeckman K, Turcksin R, Van Winkel L, Gucciardo L, Laubach M, Peersman W, Swinnen E. The experiences of last-year student midwives with High-Fidelity Perinatal Simulation training: A qualitative descriptive study. Women Birth. 2017 Jun;30(3):253-261. doi: 10.1016/j.wombi.2017.02.014. Epub 2017 Mar 22. PMID 28341585
- [Result] Walker S, Breslin E, Scamell M, Parker P. Effectiveness of vaginal breech birth training strategies: An integrative review of the literature. Birth. 2017 Jun;44(2):101-109. doi: 10.1111/birt.12280. Epub 2017 Feb 17. PMID 28211102
- [Result] Walker S, Reading C, Silverwood-Cope O, Cochrane V. Physiological breech birth. Evaluation of a training programme for birth professionals. Pract Midwife. 2017 Feb;20(2):25-8. PMID 30462429